CLINICAL TRIAL: NCT01482000
Title: Detection and Intervention on Mild/Moderate Chronic Obstructive Pulmonary Disease by Traditional Chinese Medicine Treatment and Application
Brief Title: Does Pulmonary Daoyin of China Give Additional Benefit Over Usual Therapy in Management of Stable Chronic Obstructive Pulmonary Disease?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daoyin therapy for COPD
Record Dates: First submitted 2011-11-18; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Adult; therapeutic use; Humans; Treatment Outcome; daoyin therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary daoyin therapy of China (Experimental): The intervention group will perform a 3 months pulmonary daoyin of China therapy program which consists of training and patient education. They will be evaluated with some tests for the study.
  Interventions: Other: Pulmonary daoyin therapy of China
- Control (Active Comparator): The control group will get the usual care with some additional tests for the study.
  Interventions: Other: usual care

INTERVENTIONS:
Other: Pulmonary daoyin therapy of China — The intervention group will perform a 3 months pulmonary daoyin of China therapy program which consists of training and patient education. They will be evaluated with some tests for the study.
  Arms: Pulmonary daoyin therapy of China
Other: usual care — The control group will get the usual care with some additional tests for the study.
  Arms: Control

SUMMARY:
The purpose of this study is to compare the exercise capacity and pulmonary function test parameters of Chronic Obstructive Pulmonary Disease (COPD) patients who underwent usual care with and without pulmonary daoyin therapy of China in community.

DETAILED DESCRIPTION:
This is a multicenter, randomized, none-blind, controlled study to evaluate the effect of pulmonary daoyin therapy in moderate to very severe COPD subjects. Following a 14 day run-in period, approximately 464 subjects will be randomly assigned to none-blind treatment for 3 months. The primary measure of efficacy is the Exercise Capacity (6MWD) and spirometric values (e.g. FEV1). Secondary efficacy measures include Dyspnea (MMRC), Quality of life (CAT,SF-36), frequency of exacerbations. Safety will be assessed through the collection of adverse events. There will be a total of 4 study visits (randomization, and after 1,2,3 months of treatment).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of moderate to very severe COPD.
* Age between 40 and 80 years.
* Without participation in other interventional trials in the previous one month.
* With the informed consent signed.

Exclusion Criteria:

* Patients with poor mobility that can not do the exercise, i.e. wheelchair bound.
* Pregnant or breast-feeding women.
* Resting pulmonary artery pressure > 45mmHg.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Patients with severe comorbidities, including acute myocardial infarction and unstable angina pectoris.
* Patients with post exercise syncope and osteoarthrosis that affect movement.
* Complicated with severe heart failure (class II to IV NYHA heart function).
* Complicated with bronchial asthma, bronchiectasis or active tuberculosis;
* Complicated with obliterative bronchiolitis or diffuse pantothenic bronchiolitis，
* Complicated with pneumothorax, pleural effusion or pulmonary embolism.
* Complicated with neuromuscular disorder which affects the respiration.
* Complicated with tumors .
* Complicated with serious hepatic and renal diseases.
* Long periods of bed rest .
* Participating in other trials or allergic to the used medicine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Distance Test ( 6MWD) | Change from Baseline in 6MWD at month 3 of the treatment phase
Forced expiratory volume in one second, FEV1 | Change from Baseline in FEV1 at month 3 of the treatment phase

SECONDARY OUTCOMES:
Modified Medical Research Council (MMRC) scale | Change from Baseline in MMRC at month 1, 2 and 3 months of the treatment phase
Quality of life | Change from Baseline in CAT and SF-36 at month 3 of the treatment phase
  using COPD Assessment Test (CAT) and short-form 36-item questionnaire (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Li jiansheng, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine

REFERENCES:
- [Derived] Yu XQ, Li JS, Li SY, Xie Y, Wang MH, Zhang HL, Wang HF, Wang ZW. Functional and psychosocial effects of pulmonary Daoyin on patients with COPD in China: study protocol of a multicenter randomized controlled trial. J Integr Med. 2013 Mar;11(2):140-6. doi: 10.3736/jintegrmed2013015. PMID 23506695